CLINICAL TRIAL: NCT03067272
Title: Pilot Bi-Lateral Tubal Occlusion Trial for Female Permanent Contraception
Acronym: BLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Femasys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CP-100-006
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-02

CONDITIONS: Contraception
Keywords: Permanent contraception; Birth control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FemBloc® Permanent Contraceptive System (Experimental): Treatment of women who desire permanent birth control (female sterilization) by occlusion of the fallopian tubes.
  Interventions: Device: FemBloc® Permanent Contraceptive System

INTERVENTIONS:
Device: FemBloc® Permanent Contraceptive System — The FemBloc Permanent Contraceptive System consists of treatment with a Delivery System and Biopolymer, and a confirmation test with the FemChec® Tubal Occlusion Confirmation device as part of a sonographic hysterosalpingogram (Sono HSG).

SUMMARY:
Prospective, multi-center, pilot study evaluating the safety of the FemBloc® Permanent Contraceptive System for female sterilization in preventing pregnancy.

DETAILED DESCRIPTION:
Prospective, multi-center, pilot study of subjects undergoing the FemBloc Permanent Contraceptive System procedure conducted at 5 sites in the U.S. following 49 subjects total. The objective of the trial is to evaluate the safety of the FemBloc Permanent Contraceptive System for female sterilization in preventing pregnancy through the 3-month confirmation test visit. Femasys also intends to continue follow-up of pilot subjects for safety a total duration of approximately 68 months after the FemBloc treatment procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female, 21 - 45 years of age desiring permanent birth control
* Agreement to use temporary birth control (excluding IUC) until documented occlusion
* Sexually active (minimum of 4 coital acts per month) with male partner who is not known or suspected to be sterile
* At low risk for sexually transmitted infection and / or monogamous
* Reasonably certain subject is not pregnant at time of screening and procedure visits
* Willing to accept the risk of pregnancy while relying solely on FemBloc for contraception
* Signs informed consent agreeing to the protocol requirements and is able to meet the trial schedule

Exclusion Criteria:

* Uncertainty about the desire to end fertility
* Suspected or confirmed pregnancy
* Prior tubal surgery
* Uterine anomaly such as unicornuate, bicornuate, arcuate, septate, and didelphic
* Known endometrial or myometrial conditions (e.g. submucous leiomyoma) or uterine position (e.g. retroflexion or anteflexion) that would interfere with insertion tube midline fundal placement, access to uterine cornua, or lateral deployment of the catheters
* Any condition which may prohibit proper visualization of the cervix or not allow the uterus to be appropriately instrumented
* Active or untreated pelvic infection
* Presence or suspicion of gynecologic malignancy
* Any condition or medical treatment (e.g. systemic corticosteroids or chemotherapy) that compromises immune system
* Post-partum or pregnancy termination <6 weeks of scheduled procedure
* Complicated IUC removal on the day of FemBloc treatment (e.g. use of intracavitary instrument for removal, bleeding, excessive pain)
* Scheduled to undergo concomitant intrauterine procedures at the time of FemBloc treatment or planning any uterine procedure within the 3 months after treatment
* Known hypersensitivity to cyanoacrylate or formaldehyde
* Prior history of ectopic pregnancy
* Abnormal uterine bleeding of unknown etiology
* Any general health condition or systemic disease that may represent, in the Investigator's opinion, a potential increased risk associated with device use or pregnancy, or that would not allow them to complete the trial

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects who experience an Adverse Event divided by the number of subjects exposed to the FemBloc treatment procedure | 5 months
  Evaluated up to 3 months after the FemBloc treatment procedure

OTHER OUTCOMES:
Number of subjects who experience an Adverse Event divided by the number of subjects exposed to the FemBloc Confirmation test | 5 months
  Evaluated at 3 months after the FemBloc treatment procedure
Number of subjects who experience an Adverse Event divided by the number of subjects exposed to the FemBloc Biopolymer | 5 months
  Evaluated up to 3 months after the FemBloc treatment procedure

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Sponsor Clinical Affairs
Locations (4):
- United States (4):
  - Altus Research Inc., Lake Worth, Florida
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No